CLINICAL TRIAL: NCT07042152
Title: Sensor Enhanced Activity Motivation After Stroke
Brief Title: Wearable Device and Behavioral Support for Enhancing Arm Use After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, David Reinkensmeyer, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2621
Record Dates: First submitted 2025-05-19; First posted 2025-06-27 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Stroke Patients
Keywords: Sensor; SmartWatch; Stroke Recovery; Stroke Rehabilitation; Motivational Interviewing
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement Variability (Experimental): The movement variability group will have a smartwatch app that records movement variability. Their movement goal will be centered on increasing their total movement variability as measured by the watch.
  Interventions: Other: Smartwatch App for Movement Variability; Behavioral: Motivational Interviewing (Within Subjects)
- Active Time (Control) (Placebo Comparator): This group will only receive active-time feedback (the number of minutes and hours moving the upper extremity). Their goal will focus on increasing their total movement time.
  Interventions: Other: Smartwatch App for Active Time; Behavioral: Motivational Interviewing (Within Subjects)

INTERVENTIONS:
Other: Smartwatch App for Movement Variability — This app measures movement variability in the upper extremity as described in our previous study (doi:10.3390/s24165266).
  Arms: Movement Variability
Other: Smartwatch App for Active Time — The other software we are using measures total active time of the upper extremity.
  Arms: Active Time (Control)
Behavioral: Motivational Interviewing (Within Subjects) — Motivational Interviewing is an established therapeutic technique designed to increase patient adherence to therapy by addressing ambivalence. The motivational Interviewing sessions will include a variety of techniques such as: Open ended questions, Active Listening, Affirmation, Summarization, Questions focused on change talk, and Providing Information.

SUMMARY:
The goal of this study is to determine the effectiveness of behavioral support and feedback from a wearable device that senses arm movement in improving upper extremity function in a pilot, randomized controlled trial with chronic stroke patients

DETAILED DESCRIPTION:
In this randomized controlled trial, the investigators will evaluate two telerehabilitation strategies for increasing arm use at home: a smartwatch app and a psychological intervention. The psychological intervention aims to address ambivalence and enhance motivation, while the smartwatch provides feedback on arm movement variability. The investigators hypothesize that combining the psychological intervention with smartwatch feedback will lead to greater improvements in arm use and upper extremity recovery

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age
* Experienced a single or multiple, ischemic or hemorrhagic stroke, with unilateral weakness, over six months previously
* An ability to score at least 3 blocks on the Box and Block Test. BBT score of the affected arm is at least 5% worse than that present with the unaffected arm.
* Absence of major depression, as defined by DSM V criteria or a score on the Geriatric Depression Scale < 10.

Exclusion Criteria:

* Any substantial decrease in alertness, language reception, or attention
* Single or multiple, ischemic or hemorrhagic stroke less than 6 months ago
* Severe muscle tone at the upper extremity (score ≥ 3 on the Modified Ashworth Spasticity scale)
* Pregnant or lactating
* Advanced liver, kidney, cardiac, or pulmonary disease
* Coexistent major neurological disease
* Coexistent major psychiatric disease
* Plans to alter any current participation in other rehabilitation therapy in the time period of the study
* A terminal medical diagnosis consistent with survival < 1 year
* A history of significant alcohol or drug abuse in the prior 3 years
* Current enrollment in another study related to stroke or stroke recovery
* Any other medical contraindication to participation in the study, as evaluated by our team physician.
* Visual Analog of Pain Scale Score of 7 or greater

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Variability Measurement | From enrollment to the end of treatment and follow up measurement (9 weeks)
  The amount of variability for the impaired upper extremity will be quantified by the variety of movements performed.

SECONDARY OUTCOMES:
Active Time | From enrollment to the end of treatment and follow up measurement (9 weeks)
  This outcome measures the active time of the impaired upper extremity in minutes and hours.
Fugl-Meyer Arm Motor Assessment | Initial Visit, First follow up, Second follow up
  The Fugl-Meyer Arm Motor Assessment measures motor impairment, movement coordination, reflexes, and functional ability of the upper limb in stroke patients, providing a quantitative evaluation of motor recovery based on a standardized scoring system.
Box and Blocks Test | Initial Visit, First follow up, second follow up
  The Box and Blocks Test (BBT) measures manual dexterity, unilateral gross motor function, and upper limb coordination in stroke patients by assessing the number of blocks transferred within a set time, providing an objective indicator of motor recovery and functional hand use.
Nine Hole Peg Test | Initial Visit, First follow up, Second follow up
  The 9-Hole Peg Test (9HPT) measures fine motor coordination, dexterity, and finger-hand function by assessing the speed at which a participant can place and remove pegs from a board.
Motor Activity Log (MAL) | Initial Visit, First follow up, Second follow up
  The Motor Activity Log (MAL) measures the amount and quality of spontaneous arm use in daily activities in stroke patients with hemiparesis, using patient-reported ratings on a structured questionnaire to assess real-world upper limb function.
Open Point | Initial Visit, First follow up, Second follow up
  Open Point measures proprioception in patients with impaired upper extremity function due to stroke.
  Cornella-Barba, G., Farrens, A. J., Johnson, C. A., Garcia-Fernandez, L., Chan, V., & Reinkensmeyer, D. J. (2024). Using a Webcam to Assess Upper Extremity Proprioception: Experimental Validation and Application to Persons Post Stroke. Sensors (Basel, Switzerland), 24(23), 7434. https://doi.org/10.3390/s24237434
NIH Stroke Scale | Initial Visit, First follow up, Second follow up
  The NIH Stroke Scale (NIHSS) measures stroke severity by assessing neurological function, including consciousness, motor and sensory abilities, language, vision, and inattention to quantify impairment.
Fatigue Severity Scale (FSS) | Initial Visit, First follow up, Second follow up
  The Fatigue Severity Scale (FSS) measures the impact of fatigue on daily functioning and quality of life, assessing both the severity and the effect of fatigue on physical and cognitive activities through a self-reported questionnaire.
Fugl-Meyer Sensory Assessment: Touch and Proprioception | Initial Visit, First follow up, Second follow up
  The Fugl-Meyer Sensory Assessment evaluates sensory function in stroke patients by assessing light touch sensitivity and joint position sense (proprioception) in the affected limbs.
Kinect: Sensor-based Upper Extremity Reachable Workspace Evaluation | Initial Visit, First follow up, Second follow up
  The Kinect workspace measures the three-dimensional reachable space of the upper limb in hemiplegic stroke patients by tracking movement using a Kinect sensor, providing an objective assessment of functional reaching ability.
  Lee, Y. M., Lee, S., Uhm, K. E., Kurillo, G., Han, J. J., & Lee, J. (2020). Upper Limb Three-Dimensional Reachable Workspace Analysis Using the Kinect Sensor in Hemiplegic Stroke Patients: A Cross-Sectional Observational Study. American journal of physical medicine & rehabilitation, 99(5), 397-403. https://doi.org/10.1097/PHM.0000000000001350

OTHER OUTCOMES:
Geriatric Depression Scale | Initial Visit, First follow up, Second follow up
  The Geriatric Depression Scale (GDS) is a screening tool designed to assess depressive symptoms in older adults.
Intrinsic Motivation Inventory (IMI) | Initial Visit, First follow up, Second follow up
  The Intrinsic Motivation Inventory (IMI) measures a person's subjective experience of motivation in a given activity, assessing factors such as interest/enjoyment, perceived competence, effort, value/usefulness, and relatedness through a self-report questionnaire.
Modified Ashworth Spasticity Scale | Initial Visit, First follow up, Second follow up
  The Modified Ashworth Spasticity Scale measures muscle spasticity by assessing resistance to passive movement in a limb, grading it on a scale from 0 (no increase in tone) to 4 (rigid in flexion or extension).
Visual Analog of Pain Scale | Initial Visit, First follow up, Second follow up
  Rating Pain on a scale of 1-10.
Montreal Cognitive Assessment | Initial Visit, First follow up, Second follow up
  The Montreal Cognitive Assessment (MoCA) is a screening tool that evaluates cognitive function by assessing domains such as memory, attention, language, visuospatial skills, and executive function to detect mild cognitive impairment.
System Usability Scale | second visit
  System Usability Scale is a short questionnaire that asks about your experience using a device or system.

CONTACTS AND LOCATIONS:
Overall Officials: David Reinkensmeyer, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share Individual Participant Data (IPD) with external researchers to ensure compliance with UCI's data management requirements, maintain participant confidentiality, and restrict access to approved UCI researchers using only deidentified data within our institution

REFERENCES:
- [Background] Schwerz de Lucena D, Rowe JB, Okita S, Chan V, Cramer SC, Reinkensmeyer DJ. Providing Real-Time Wearable Feedback to Increase Hand Use after Stroke: A Randomized, Controlled Trial. Sensors (Basel). 2022 Sep 14;22(18):6938. doi: 10.3390/s22186938. PMID 36146287